CLINICAL TRIAL: NCT05115565
Title: The Effect of Transcutaneous Electrical Nerve Stimulation on Pain, Functionality and Quality of Life in Patients With Total Knee Replacement
Brief Title: The Effects of Transcutaneous Electrical Nerve Stimulation in Patients With Total Knee Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Nilgun Ozbas, Assistant Professor, Bozok University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2017-KAEK-189_2021.09.22_05
Record Dates: First submitted 2021-09-05; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Total Knee Replacement; Transcutaneous Electrical Nerve Stimulation; Total Knee Replacement Surgery
Keywords: Total knee replacement; Transcutaneous Electrical Nerve Stimulation; Pain; Nursing; Quality of life
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the study, patients will not be left blind. The assignment to the groups will be carried out by an independent researcher, and the group will be notified via telephone after the practitioner researcher has approved, evaluated the criteria and performed the pre-tests. At the same time, groups will be named A and B and researchers will be blinded during statistical analysis and reporting.The questionnaires to be applied to the patients included in the study will be administered by an independent researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): When the patients are admitted to the clinic, the patient identification form and the SF-36 Quality of Life Scale will be filled by face-to-face interview method. On the morning of the operation, before the operation, the GCS, EHA and WOMAC index will be filled. After the operation, the pain during rest and movement (24., 48., 72., 96. hours and 15. days) will be evaluated with VAS. The total amount of analgesics used by the patients will be recorded by looking at the nurse observation form records where the nurses recorded the drugs they administered at the 24th, 48th, 72nd, and 96th hours after the surgery, and by asking the patients on the 15th day after discharge. The WOMAC Index will be re-administered at discharge and on the 15th day, and the VCS, ROM, and the SF-36 Quality of Life Scale on the 15th day.
- Intervention group (Experimental): Unlike the control group, the patients in the intervention group will be informed about TENS and the application will be made. The electrodes of TENS will be placed 2 cm below and 2 cm above the incision site. TENS settings Frequency: 100 Hz; Pulse width (duration): 150 μs; Flow Intensity (Amplitude): By adjusting it to be 30 mA, TENS will be applied 3 times a day (09.00, 13.00, 17.00) for 20 minutes during the time the patients stay in the clinic (3 days).It is planned to start the TENS application the day after the surgery.
  Interventions: Device: TENS (Transcutaneous Electrical Nerve Stimulation) Application

INTERVENTIONS:
Device: TENS (Transcutaneous Electrical Nerve Stimulation) Application — Conventional (traditional) TENS will be applied to the patients. The frequency will be 100 Hz, the pulse width (time) will be 150 μs, the current intensity (amplitude) will be 30 mA. In addition to routine care and treatment, TENS will be applied to intervention group patients.
  Arms: Intervention group

SUMMARY:
Total Knee Replacement (TDP) is considered the best treatment option available when conservative methods such as anti-inflammatory or physical therapy fail. However, TDP surgeries are also a serious trauma that causes severe pain in patients. Uncontrollable pain exacerbates the stress response and causes morbidity and mortality by causing negative changes in the neuroendocrine, respiratory, cardiovascular, gastrointestinal, renal and immune systems. Therefore, the relief of pain has very important effects on the patient's recovery process, functional status and quality of life. Transcutaneous Electrical Nerve Stimulation (TENS) is one of the non-pharmacological methods for pain relief in TDP surgeries. This study was planned as a randomized controlled trial to examine the effects of TENS after TDP on acute pain, functionality and quality of life.

DETAILED DESCRIPTION:
Nowadays, it is seen that the results of an increasing number of TDP surgeries increase patient satisfaction and have satisfactory results. However, TDP surgery is a serious trauma that causes pain in patients.

TENS is an easy-to-apply, inexpensive, noninvasive, noninvasive method that uses electrical current to activate nerves with therapeutic effects in the treatment of acute and chronic pain. It is also seen as a promising practice in patients undergoing total knee replacement surgery by the American Society of Regional Anesthesia and Pain Medicine (ASRA) and the European Society of Regional Anaesthesia and Pain Therapy (ESRA).

The study was planned as a randomized controlled study to examine the effect of TENS on acute pain, functionality and quality of life after TDP. The hypotheses of the study; H1a- TENS applied after TDP positively affects the level of pain in patients. H1b- TENS applied after TDP affects the improvement in functional status in patients.

H1c- TENS applied after TDP reduces the analgesia consumption of patients. H1d- TENS applied after TDP positively affects the quality of life of patients. Type of Study: Randomized controlled trial. Method: 52 patients (26 controls, 26 interventions) who underwent total knee replacement surgery will be randomized and divided into two groups as intervention and control groups. TENS will be applied to the intervention group in addition to the routine treatment and care in the clinic, on the other hand, no intervention will be made to the control group other than routine treatment and care. Data will be collected with Patient identification form, Pain Evaluation Form, Visual Analogue Scale (VAS), Analgesic Drug Tracking Form, Joint Range of Motion (ROM) Follow-up Form, Western Ontario and McMaster Universities Arthritis Index (WOMAC), Quality of Life Scale (SF-36).

While evaluating the data, it is planned to be analyzed as randomized.It is planned to use multiple completion methods when there are missing data.Statistical analyzes are planned to be evaluated with the SPSS-24 package program. It is planned to use frequency charts and descriptive statistics in order to interpret the data, parametric techniques for normal distributions and non-parametric techniques for non-normal distributions.

ELIGIBILITY:
Inclusion Criteria:

* Not have had knee replacement surgery before,
* Having unilateral prosthesis surgery,
* Not having a pacemaker or arrhythmia,
* Not having neurological deficit,
* Absence of sensory loss, paresthesia or hyporeflexia,
* Not having local or systemic infection,
* Not using opioids or TENS before surgery,
* Not having history of chronic pain,
* Not having history of alcohol or drug use,
* Not having a psychiatric history,
* Not having been done to apply epidural analgesia in the postoperative period,
* Not having serious complications after surgery,
* Not having a history of neurological disease (SVO, epilepsy, dementia, etc.),
* Not having active tumor or cancer,
* Not having fractures or dislocations,
* Absence of signs of venous thromboembolism,
* Having an ASA score of I and II,
* Agree to participate in the research and
* Know how to read and write

Exclusion Criteria:

* Undergoing previous knee replacement surgery,
* Having double-sided prosthesis surgery,
* Having a pacemaker and arrhythmia,
* Having a neurological deficit,
* Having loss of sensation, paresthesia or hyporeflexia,
* Having local or systemic infection,
* Having been used opioids and or TENS before surgery,
* Having a history of chronic pain,
* Having a history of alcohol or drug use,
* Having a psychiatric history,
* Administering epidural analgesia in the postoperative period,
* Developing serious complications after surgery,
* Having a history of neurological disease (SVO, epilepsy, dementia, etc.),
* Having an active tumor or cancer,
* Having fracture or dislocation,
* Having symptoms of venous thrombosis,
* Not having ASA score I or II,
* Not agreeing to participate in the study,
* Illiteracy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-11-15 (Estimated); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) Change | 1st day of admission to the clinic change VAS score at before intervention, 24th postoperative hour change from baseline VAS score before the intervention, postoperative 48th, 72th and 96th hours,15th day change from baseline VAS score after intervention
  The Visual Analogue Scale (VAS) is a scale where the pain is evaluated between 0-10 (0; no pain, 10; unbearable pain) on a ruler that can be used horizontally or vertically, on which the patient can mark his or her own pain.The length of the distance from the point where there is no pain to the point marked by the patient is measured in centimeters and the numerical value found shows the severity of the patient's pain. It is used in various populations, including patients with total knee replacement, to evaluate both the severity of pain and the effectiveness of treatment/intervention on pain.

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index (WOMAC) Change | 1st day of admission to the clinic change WOMAC score at before intervention, change from baseline the WOMAC score at 4th postoperative day, 15th postoperative day change from baseline WOMAC score
  WOMAC is planned to be used to assess functionality in patients.The score to be taken from the scale is between 0-100. An increase in score indicates deterioration in physical function.
  The WOMAC index is a valid and reliable index that is widely used for the evaluation of patients with osteoarthritis. The index consists of three parts and 24 questions in which pain, stiffness and physical function are questioned. Each question was scored according to the Likert scale as 0=absent, 1=mild, 2=moderate, 3=severe, 4=very severe. The score of each section is calculated in itself and the total score varies between 0 and 100. High scores indicate an increase in pain and stiffness, and deterioration in physical function.
The Quality of Life Scale (SF-36) Change | 1st day of admission to the clinic change quality of life score at before intervention, 15th postoperative day change from baseline quality of life score
  The Quality of Life Scale (SF-36), one of the most used scales to measure quality of life; It is a self-assessment scale that can be filled in a short time and is highly sensitive.While applying the scale, individuals are asked to answer considering the last 4 weeks. The scale consists of 36 questions and 8 sub-parameters (body pain, limitation due to physical problems, limitation due to mental problems, mental well-being, fatigue, general health perception, social function and physical function). In scoring, each parameter is evaluated between 0 and 100 points. A score of 0 indicates poor health, and a score of 100 indicates good health. The higher the score, the higher the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Nilgün Özbaş, Assist. Prof, Principal Investigator — Bozok University; Emre Ersoy, Assist. Prof, Study Chair — Bozok University; Hacı Ali Olçar, Doctor, Study Chair — Bozok University
Locations (1):
- Yozgat Bozok University Research and Application Hospital, Yozgat, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No